CLINICAL TRIAL: NCT04664946
Title: Intra-arterial Neuroprotective Strategy for Ischemic STroke Patients With No Reperfusion Therapy (INSIST-NRT): One Single Center, Safety and Feasibility Study
Brief Title: Intra-arterial Neuroprotective Strategy for Ischemic STroke Patients With No Reperfusion Therapy (INSIST-NRT)
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Hui-Sheng Chen (Other)
Responsible Party: Sponsor-Investigator, Hui-Sheng Chen, Director, General Hospital of Shenyang Military Region
Organization: General Hospital of Shenyang Military Region (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: k（2020）31
Record Dates: First submitted 2020-11-30; First posted 2020-12-11 (Actual); Last update posted 2025-08-21 (Actual); Status verified 2025-08

CONDITIONS: Ischemic Stroke; Neuroprotection
MeSH Terms: conditions — Ischemic Stroke

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Intra-arterial administration of 3-n-butylphthalide (Experimental): Intra-arterial administration of 3-n-butylphthalide for 24 hours via microcatheter at 17.36 ug/min.
  Interventions: Drug: Intra-arterial administration of neuroprotective agents

INTERVENTIONS:
Drug: Intra-arterial administration of neuroprotective agents — Intra-arterial administration of 3-n-butylphthalide for 24 hours via microcatheter at 17.36 ug/min.

SUMMARY:
To explore the safety and feasibility of intra-arterial neuroprotective strategy in acute ischemic stroke patients who missed recanalization operation.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥18 years;
2. Major neurologic deficits: 6≤NIHSS≤20;
3. Missing recanalization therapy (IVT or EVT) or progressive stroke, which was defined as symptoms worsen in 48 hours (an increase in NIHSS more than 4);
4. Premorbid mRS 0 or 1;
5. Signed informed consent.

Exclusion Criteria:

1. Modified Rankin Score >2 caused by a history of prior stroke;
2. Patients who underwent intravenous thrombolysis or Endovascular treatment;
3. Coagulation disorders, systematic hemorrhagic tendency, thrombocytopenia （ <80000/mm3;
4. Severe hepatic or renal dysfunction, increase in ALT or AST (more than 2 times of upper limit of normal value), increase in serum creatinine (more than 1.5 times of upper limit of normal value) or requiring dialysis;
5. Severe hypertension (systolic blood pressure over 200mmHg or diastolic blood pressure over 110 mmHg);
6. Unsuitable for this clinical studies assessed by researcher.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2020-12-01 (Actual); Primary Completion 2026-05-01 (Estimated); Study Completion 2026-05-01 (Estimated)

PRIMARY OUTCOMES:
Proportion of server adverse events | 48 hours
  server adverse events including femoral artery dissection, local thrombosis, seudoaneurysm, arteriovenousfistula, etc.

SECONDARY OUTCOMES:
Proportion of patients with modified Rankin Score 0 to 1 | 90 days
  Proportion of patients with modified Rankin Score 0 to 1
Proportion of patients with modified Rankin Score 0 to 2 | 90 days
  Proportion of patients with modified Rankin Score 0 to 2
Modified Rankin Score | 90 days
  Modified Rankin Score
Decrease in national institutes of health stroke scale (NIHSS) | 48 hours
  Decrease in NIHSS scoring at 48 hours after the treatment
Proportion of symptomatic intracranial hemorrhage (sICH) | 48 hours
  sICH was defined as 4 or more increase in NIHSS caused by hemorrhage
Proportion of intraparenchymal hemorrhage (PH1 and PH2) | 48 hours
  Proportion of intraparenchymal hemorrhage (PH1 and PH2) within 48 hours after the treatment
Changes in cerebral edema | 48 hours
  Cerebral edema was determined by cerebral volume or midline shift
All causes of death within 48 hours after the treatment | 48 hours
  All causes of death within 48 hours after the treatment
Differences in serum factors levels in different artery region | 0 hour
  Differences in serum factors levels in different Bessel region before recanalization

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Neurology, General Hospital of Northern Theater Command, Shenyang, China